CLINICAL TRIAL: NCT00590993
Title: Magnetic Resonance Imaging and Spectroscopy of the Prostate
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-136
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: MRSI; MRI; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 - MRSI / MRI
  Interventions: Other: MRI and MRSI

INTERVENTIONS:
Other: MRI and MRSI — Compare treatment impact when using MRI and MRSI

SUMMARY:
Past studies have shown that MRI is useful for staging prostate cancer. This study will use magnetic resonance spectroscopic imaging (MRSI) to obtain more information. MRSIs with MRIs help doctors locate prostate cancer and determine the extent of tumor before deciding on treatment. This study looks at structural and chemical properties of prostates in prostate cancer patients before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer patients willing to undergo a MRI and MRSI exam

Exclusion Criteria:

* patients with prostate cancer and bone or lymph node metastasis
* patients who can not have an MRI exam

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology and Radiology prostate cancer patients seen at Memorial Sloan-Kettering Cancer Center
Sampling Method: Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2000-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Determine added value in combining MRSI and MRI in prostate cancer treatment | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hedvig Hricak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org